CLINICAL TRIAL: NCT00046618
Title: Mapping Novel Disease Genes for Dilated Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1187; R01HL071225 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Cardiomyopathy, Congestive; Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiovascular Diseases; Heart Diseases; Heart Failure

SUMMARY:
To identify new dilated cardiomyopathy genes by genetic linkage and mutational analyses.

DETAILED DESCRIPTION:
BACKGROUND:

Dilated cardiomyopathy (DCM) is a heritable, genetically heterogeneous disorder causing congestive heart failure. Current medical therapy has minimal impact on prognosis and cardiac transplantation is the only definitive treatment for end-stage disease. The molecular and cellular mechanisms underlying DCM are poorly defined, but the importance of single gene defects in disease pathogenesis is becoming increasingly apparent.

DESIGN NARRATIVE:

The genetic epidemiology study will identify novel dilated cardiomyopathy genes using genetic linkage and mutational analyses. The first aim is to determine the chromosomal location of novel familial dilated cardiomyopathy genes. This will be accomplished by genome-wide genotyping and genetic linkage analyses in three large families with autosomal dominant dilated cardiomyopathy. Previously identified dilated cardiomyopathy genes have been excluded in these families. The second aim is to identify mutations in novel genes that cause familial dilated cardiomyopathy by linkage and sequence analyses of candidate genes mapping to dilated cardiomyopathy loci. Once novel genes for familial dilated cardiomyopathy are identified, the third aim will be to determine the role of these genes in a large cohort of unrelated patients with familial and sporadic dilated cardiomyopathy. High throughput DNA sequence analyses will be performed to identify additional inherited and de novo mutations.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson — Mayo Clinic

REFERENCES:
- [Background] Olson TM, Michels VV, Ballew JD, Reyna SP, Karst ML, Herron KJ, Horton SC, Rodeheffer RJ, Anderson JL. Sodium channel mutations and susceptibility to heart failure and atrial fibrillation. JAMA. 2005 Jan 26;293(4):447-54. doi: 10.1001/jama.293.4.447. PMID 15671429